CLINICAL TRIAL: NCT00613275
Title: Patient Navigation in the Safety Net:CONNECTeDD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Battaglia, Tracy, Assistant Professor, Boston Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: U01CA116892-03 (NIH); U01CA116892 (NIH)
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer; Cervical Cancer
Keywords: PNRP; Navigation; Navigator; Activation; Disparities; Primary Care; Racial and Ethnic Minorities
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: patient Navigation — Assigning a patient navigator to patients with abnormal breast and cervical cancer screening results at one of 6 affiliated community health centers

SUMMARY:
The Boston University Medical Center, funded by the National Cancer Institutes will train health workers at six of its affiliated Community Health Centers to guide patients through the cancer care system. The project will help to teach patients how to communicate more effectively with their health care team in order to understand the treatment options available to them. Although not widely available, it is believed patient navigation programs are beneficial.

This research study will evaluate how well this tool works, especially among those who experience disparities in health care. The goal is to determine if having a trained navigator shortens the time between an abnormal test result and a definitive diagnosis and between a definitive diagnosis and completion of treatment for breast and Cervical cancer patients. The project also will evaluate whether navigation improves the ability to communicate with the doctor, satisfaction with patient's care and quality of life.

DETAILED DESCRIPTION:
Racial and ethnic minority groups and low-income persons experience significantly higher cancer mortality rates than other Americans. These disparities are due to at least two factors: (1) delays in follow-up of abnormal cancer screening results and (2) suboptimal management of diagnosed cancer. Patient navigation represents a promising means for addressing disparities by improving cancer related management for minority and other underserved populations. However, patient navigation for cancer has yet to be evaluated through a well-designed randomized controlled trial. Furthermore, patient navigation is likely to prove most effective and sustainable when it is integrated into primary care and helps patients be more active in their care. This combination of patient empowerment and engagement is referred to as "activation." The aim of this project is to evaluate the effectiveness and costs of such a program in a rigorous manner so that the results can be generalized and the program can be widely disseminated and implemented. We will develop, implement, and evaluate a primary care-based, patient navigation-activation program using specially-trained patient Navigators who work within one of the six affiliated Community Health Centers. We propose to investigate the effect of this intervention on timing and quality of cancer-related care. Secondary aims examine the impact of navigation on disparities in care, improvement in patient activation, and total costs. Project findings will inform national policy regarding patient navigation for cancer.

ELIGIBILITY:
Inclusion Criteria:

* Receive care at one of the 6 participating community Health centers
* Have received a positive breast or colorectal cancer screening test requiring follow-up on a different day
* Have been newly diagnosed with breast or colorectal cancer
* Have received notification by the provider of an abnormal breast or colorectal screening result

Exclusion Criteria:

* Cognitively impaired
* Institutionalized (nursing home, incarcerated)
* Children <18
* Actively involved in cancer treatment at time of presentation
* Currently or previously navigated with (a) navigation documented in the medical record or (b) patient can articulate that they are in a navigation program or case management program for cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4038 (Actual)
Dates: Start 2005-07; Primary Completion 2010-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Develop,implement and evaluate a primary care-based,patient navigation program using patient navigators in the Community Health Centers. We will investigate the effect of this intervention on timing and quality of cancer-related care | 4 years

SECONDARY OUTCOMES:
Secondary aims examine the impact of navigation on disparities in care, improvement in patient activation and total costs | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Freund, MD, MPH, Principal Investigator — Boston Medical Center; Tracy Battaglia, MD, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Battaglia TA, Darnell JS, Ko N, Snyder F, Paskett ED, Wells KJ, Whitley EM, Griggs JJ, Karnad A, Young H, Warren-Mears V, Simon MA, Calhoun E. The impact of patient navigation on the delivery of diagnostic breast cancer care in the National Patient Navigation Research Program: a prospective meta-analysis. Breast Cancer Res Treat. 2016 Aug;158(3):523-34. doi: 10.1007/s10549-016-3887-8. Epub 2016 Jul 18. PMID 27432417
- [Derived] Wells KJ, Winters PC, Jean-Pierre P, Warren-Mears V, Post D, Van Duyn MA, Fiscella K, Darnell J, Freund KM; Patient Navigation Research Program Investigators. Effect of patient navigation on satisfaction with cancer-related care. Support Care Cancer. 2016 Apr;24(4):1729-53. doi: 10.1007/s00520-015-2946-8. Epub 2015 Oct 5. PMID 26438146
- [Derived] Rodday AM, Parsons SK, Snyder F, Simon MA, Llanos AA, Warren-Mears V, Dudley D, Lee JH, Patierno SR, Markossian TW, Sanders M, Whitley EM, Freund KM. Impact of patient navigation in eliminating economic disparities in cancer care. Cancer. 2015 Nov 15;121(22):4025-34. doi: 10.1002/cncr.29612. Epub 2015 Sep 8. PMID 26348120
- [Derived] Ko NY, Darnell JS, Calhoun E, Freund KM, Wells KJ, Shapiro CL, Dudley DJ, Patierno SR, Fiscella K, Raich P, Battaglia TA. Can patient navigation improve receipt of recommended breast cancer care? Evidence from the National Patient Navigation Research Program. J Clin Oncol. 2014 Sep 1;32(25):2758-64. doi: 10.1200/JCO.2013.53.6037. Epub 2014 Jul 28. PMID 25071111